CLINICAL TRIAL: NCT05654077
Title: To Investigate the Safety and Preliminary Efficacy of EBV CAR-T Cells in the Treatment of Relapsed/Refractory EBV-positive Nasopharyngeal Carcinoma
Brief Title: EBV CAR-T Cells for Nasopharyngeal Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Guangzhou Bioresette Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-EB-10
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: CAR-T; nasopharyngeal carcinoma; Recurrent/refractory nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Immunotherapy, Adoptive; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Cell Injection (Experimental): A total of 24 patients with recurrent or refractory NPC received a single intravenous infusion of CAR-T cells at doses of 3.0 × 10^6cells/kg, 9.0 × 10^6cells/kg, and 1.5 × 10^7cells/kg, respectively, and were enrolled according to the conventional "3+3" dose escalation.
  Interventions: Biological: CAR-T Cell Injection; Drug: Fludarabine; Drug: cyclophosphamide

INTERVENTIONS:
Biological: CAR-T Cell Injection — intravenously once, and the dose group was 3.0 × 10^6cells/kg、9.0 × 10^6cells/kg、1.5 × 10^7cells/kg。
Drug: Fludarabine — Fludarabine 25~30mg/m2/d was infused intravenously for 3 consecutive days. (- 5 days to - 3 days)
  Other Names: FLUDARA
Drug: cyclophosphamide — 250~350mg/m2/d cyclophosphamide was infused intravenously for 3 consecutive days. (- 5 days to - 3 days)
  Other Names: Cytoxan

SUMMARY:
The aim of this study is to investigate the safety and preliminary efficacy of EBV CAR-T cells in the treatment of relapsed/refractory NPC

DETAILED DESCRIPTION:
The investigators designed a single-arm, open-label, "3+3" dose-escalation exploratory study. According to the subject and dose escalation test, the maximum dose or the best effective dose was determined to verify the safe and effective number of cells per body weight. A "3+3" dose escalation design was used to set three dose groups of gradually increasing CAR-T cells for therapeutic evaluation. The dose groups were 3.0×10^6cells/kg, 9.0×10^6cells/kg and 1.5×10^7cells/kg, respectively. Cell reinfusion will take place on day 0 (d0) and each subject will be observed for at least 4 weeks after receiving cell reinfusion (DLT observation period).

ELIGIBILITY:
Inclusion Criteria:

* 1)Voluntarily sign written informed consent;
* 2)Age ≥18, ≤75 years old, male and female;
* 3 )Estimated survival ≥ 3 months;
* 4) ECOG physical fitness score was 0-2;
* 5) EBV positive nasopharyngeal carcinoma was diagnosed;
* 6) Positive target detection;
* 7) At least one measurable lesion according to RECIST V1.1 solid tumor evaluation criteria;
* 8) Patients with recurrent/metastatic nasopharyngeal carcinoma who had previously failed second-line or higher systemic therapy;
* 9) Monopheresis or venous blood collection venous access can be established, and there are no other contraindications for blood cell separation;
* 10) Full organ and bone marrow function,
* 11) Toxicity and side effects left by previous anti-tumor therapy (radiotherapy, chemotherapy, targeted therapy, etc.) ≤ grade 1 (CTCAE 5.0);
* 12) Fertile subjects (male or female) must use effective medical contraception during the study period and for 6 months after the end of administration. In female subjects of reproductive age, a negative pregnancy test should be performed within 72 h prior to the first dose.

Exclusion Criteria:

* 1) There are active CNS metastases (except those stabilized by treatment);
* 2)HIV positive, HBsAg positive, HBV DNA copy number positive (quantitative test ≥1000cps/ mL), HCV antibody positive and HCV RNA positive;
* 3) Those with mental or psychological diseases who cannot cooperate with treatment and efficacy evaluation;
* 4) subjects with severe autoimmune diseases and long-term use of immunosuppressants;
* 5) Within 14 days prior to enrollment, there were active or uncontrollable infections requiring systemic treatment;
* 6) Any unstable systemic disease
* 7) Complicated with lung, brain, kidney and other important organ dysfunction;
* 8) Subjects have undergone major surgery or trauma in the 4 weeks prior to receiving cell therapy, or are expected to undergo major surgery during the study period;
* 9) Subjects received their last radiotherapy or anti-tumor therapy (chemotherapy, targeted therapy, or immunotherapy) within 4 weeks prior to receiving cell therapy;
* 10) The subject currently has or has had other malignancies that cannot be cured within 3 years, except cervical carcinoma in situ or basal cell carcinoma of the skin, and other malignancies with disease-free survival of more than 5 years;
* 11) T cells modified with chimeric antigen receptor (CAR T, TCR-T) within six months;
* 12) Combined graft versus host disease (GVHD);
* 13) Subjects who were receiving systemic steroids prior to screening and determined by the investigator to require long-term systemic steroid use during treatment (other than inhalation or topical use); And subjects who were treated with systemic steroids (except for inhalation or topical use) within 72 h prior to cell infusion;
* 14) A history of severe allergies or allergies;
* 15) Subjects requiring anticoagulant therapy;
* 16) Women who are pregnant or breast-feeding, or have a pregnancy plan within six months (for both men and women);
* 17) Researchers believe that there are other reasons not to include patients in the treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | From day 0 to day 28
  Adverse events related to cell therapy were observed on 28 days after CAR-T cell injection , as specified in the protocol

SECONDARY OUTCOMES:
Cmax | 12 months
  The amplification of CAR-T cells in peripheral blood peaked after administration
Tmax | 12 months
  Number of days of peak CAR-T cell expansion after administration
AUC(Day 0 to Day 28) | From day 0 to day 28
  The area under the curve of CAR-T cells from day 0 to day 28 after administration was plotted by the visit time of CAR-T cells in peripheral blood
ORR | 12 months
  Proportion of patients who achieved pre-defined tumor volume change and maintained the minimum time limit.Imaging examination was performed after administration, and RECIST1.1 evaluation criteria was used for evaluation
PFS | 12 months
  The time from the onset of leukocyte apheresis to the appearance of tumor progression or death
OS OS | 12 months
  The time between leukocyte apheresis and death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China